CLINICAL TRIAL: NCT00080743
Title: ZD1839 (IRESSA) In Tamoxifen-Resistant Metastatic Breast Cancer
Brief Title: Gefitinib With or Without Tamoxifen in Treating Patients With Tamoxifen-Resistant Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Norris Cotton Cancer Center (Other)
Responsible Party: Gary N. Schwartz, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000355145; DMS-0236; ZENECA-IRUSIRES0162
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Tamoxifen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamoxifen (Active Comparator): Tamoxifen 20 mg po once daily
  Interventions: Drug: gefitinib; Drug: tamoxifen citrate
- Placebo (Placebo Comparator): Placebo comparator one tablet po once daily
  Interventions: Drug: gefitinib; Drug: Placebo

INTERVENTIONS:
Drug: gefitinib — 250 mg po once daily
  Other Names: ZD1839, Iressa
Drug: tamoxifen citrate — 20 mg po once daily
  Other Names: Nolvadex
  Arms: Tamoxifen
Drug: Placebo — One pill po once daily
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Hormone therapy using tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. Combining gefitinib with tamoxifen may be effective in killing tumor cells that have become resistant (stopped responding) to tamoxifen.

PURPOSE: This randomized phase II trial is studying how well giving gefitinib together with tamoxifen works compared to gefitinib alone in treating patients with metastatic breast cancer that has stopped responding to tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the rate of clinical benefit in patients with tamoxifen-resistant breast cancer treated with gefitinib with or without tamoxifen.

Secondary

* Determine the toxic effects of these regimens in these patients.
* Determine whether changes in fludeoxyglucose F 18 uptake by positron emission tomography scan and changes in plasma DNA levels are indicators of an early response to gefitinib in these patients.
* Determine the pharmacokinetics of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to population (intent-to-treat population comprising all patients who receive 1 dose of treatment vs a subset of the intent-to-treat population, excluding patients with nonmeasurable/evaluable only disease). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen once daily. Beginning 14 days after the start of tamoxifen, patients receive oral gefitinib once daily.
* Arm II: Patients receive oral placebo once daily. Beginning 14 days after the start of placebo, patients receive oral gefitinib as in arm I.

In both arms, treatment continues for 26 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for 6 months.

PROJECTED ACCRUAL: A total of 46 patients (23 per treatment arm) will be accrued for this study within 23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic disease
* Initial clinical benefit from tamoxifen for metastatic disease, defined by 1 of the following:

  * Stable disease for 24 weeks or longer
  * Objective tumor response
* Documentation of clinical progression on tamoxifen within the past 6 weeks
* Hormone receptor status:

  * Estrogen or progesterone receptor positive on most recently analyzed biopsy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Pulmonary

* No clinically active interstitial lung disease

  * Patients with asymptomatic chronic stable radiographic changes are eligible

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known hypersensitivity to gefitinib
* No other malignancy within the past 5 years except basal cell carcinoma or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent trastuzumab (Herceptin®)

Chemotherapy

* No concurrent cytotoxic chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 2 weeks since other prior tamoxifen
* No concurrent hormone replacement therapy
* No other concurrent antiestrogens, including raloxifene
* No concurrent aromatase inhibitors
* No concurrent megestrol
* Concurrent systemic steroids for reasons other than skin toxicity allowed provided the steroids were initiated before study entry AND dose remains stable

Radiotherapy

* Concurrent palliative radiotherapy as short-term treatment for symptomatic bone metastases allowed provided other evaluable sites of disease are present AND treatment lasts no more than 14 days

Surgery

* Recovered from prior oncologic or other major surgery
* No concurrent surgery during and for 7 days after study treatment
* No concurrent ophthalmic surgery

Other

* Recovered from all prior therapy (except alopecia)
* More than 30 days since prior investigational drugs
* No other concurrent investigational agents
* No concurrent administration of any of the following:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
  * Systemic retinoids
  * CYP3A4 inhibitors (e.g., itraconazole)
  * Drugs that cause significant sustained elevation in gastric pH ≥ 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-01; Primary Completion 2005-04 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (complete response, partial response, and stable disease) for 26 weeks | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary N. Schwartz, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States